CLINICAL TRIAL: NCT00670306
Title: Cetrorelix Pamoate (AEZS-102) in Patients With Symptomatic BPH: an Open-Labeled Safety and Efficacy Assessment Study
Brief Title: Cetrorelix Pamoate IM Regimens in Patients With Symptomatic Benign Prostatic Hyperplasia (BPH)
Acronym: AEZS-102-Z041
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Daniel Croteau / Medical Manager, AEterna Zentaris
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEZS-102-Z041
Record Dates: First submitted 2008-04-22; First posted 2008-05-01 (Estimated); Results first posted 2011-01-19 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Benign Prostatic Hypertrophy
Keywords: Cetrorelix; BPH
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetrorelix 78 mg (Experimental): Drug: Cetrorelix 52 mg week 0, and 26 mg week 2, intra muscular-2 doses in 2 weeks and follow up to week 26.
  Interventions: Drug: Cetrorelix Pamoate

INTERVENTIONS:
Drug: Cetrorelix Pamoate — Cetrorelix Pamoate IM, 52 mg week 0, 26 mg week 2,
  Other Names: Cetrorelix pamoate, D-20762, AEZS-102

SUMMARY:
Benign Prostatic Hyperplasia (BPH) is the most common hyperplastic disease occuring in human males over the age of 50 which increases in prevalence with age and 40% of males reported moderate or severe urinary symptoms of prostatism by the age of 50 to 80. The purpose of this study is to collect safety and efficacy data for this dosage regimen of cetrorelix pamoate.

For this study, study medication (Cetrorelix pamoate) is administered by injection in the buttocks (Intramuscular).

ELIGIBILITY:
Inclusion Criteria:

* Benign Prostatic Hyperplasia, based on medical history
* Voiding symptoms
* Uroflow (max) 5-15mL/sec

Exclusion Criteria:

* Urgent need for prostate surgery
* History of allergic reaction to peptide
* Major organ dysfunction
* Prior surgical treatment of the prostate or bladder
* Current or recent treatment with sexual hormone drugs or 5 α reductase inhibitors or botulinum toxin type a (Botox) within the last 6 months prior to trial medication at Week 0 or with α blockers or saw palmetto within the last 6 weeks prior to trial medication at Week 0
* Urologic disorders including neurogenic bladder dysfunction due to diabetes mellitus or documented neurologic disorder, urethral stricture disease or history of pelvic radiation therapy
* History of acute obstructive, infectious, or neurological disorders of the genitourinary tract within the last 3 months

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (69):
- United States (56):
  - Urology Centers of Alabama, Homewood, Alabama
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - South Orange County Medical Research Center, Laguna Hills, California
  - California Professionnal Research, Newport Beach, California
  - Northern California Research, Sacramento, California
  - San Diego Uro Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - West Coast Clinical Research, Tarzana, California
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Connecticut Clincal Research Center, LLC, Middlebury, Connecticut
  - Urological Associates of Bridgeport, Trumbull, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - University Urologists, Lake Worth, Florida
  - Specialists in Urology, Naples, Florida
  - Winter Park Urology, Orlando, Florida
  - Florida Urology Specialists, Sarasota, Florida
  - Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - Welborn Clinic, Newburgh, Indiana
  - The Iowa Clinic, Des Moines, Iowa
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Bel Air, Maryland
  - Myron I. Murdock M.D. LLC, Greenbelt, Maryland
  - Michigan Institute of Urology, Troy, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Five Valleys Urology, Missoula, Montana
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Meridian Clinical Research LLC, Omaha, Nebraska
  - Sheldon J. Freedman, MD, LTD, Las Vegas, Nevada
  - Lawrenceville Urology, P.A. dba AdvanceMed Research, Lawrenceville, New Jersey
  - Delaware Valley Urology, LLC-Voorhees, Voorhees Township, New Jersey
  - Delaware Valley Urology, LLC, Woodlane, New Jersey
  - Upstate Urology, Albany, New York
  - Capital Region Urologic Surgeons, Albany, New York
  - Medical & Clinical Research Associates, Bay Shore, New York
  - Urological Surgeons of Long Island, Clinical Research Division, Garden City, New York
  - Advanced Urology, Jackson Heights, New York
  - New York University School of Medicine, New York, New York
  - University Urology Associates, New York, New York
  - Urology Associates-Rochester, Rochester, New York
  - Northeast Urology Research, Concord, North Carolina
  - Piedmont Medical Group, Winston-Salem, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Parkhurst Research Oganization Inc., Bethany, Oklahoma
  - Urologic Consultants of SEPA, Bala-Cynwyd, Pennsylvania
  - Urological Associates of Lancaster, Lancaster, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Matrix Research, Greer, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - University of Texas Southwestern Medical Center, Department of Urology, Dallas, Texas
  - Salt Lake Research, PLLC, Salt Lake City, Utah
  - Urology of Virginia, Virginia Beach, Virginia
  - Seattle Urology Research, Seattle, Washington
- Canada (13):
  - Can-Med Clinical Research Inc., Victoria, British Columbia
  - The Male / FemaleHealth and Research Center, Barrie, Ontario
  - Dr. Jonathan Giddens, Brampton, Ontario
  - Brantford Urology Research, Brantford, Ontario
  - Guelph Urology Associates, Guelph, Ontario
  - Urologic Associates, Urologic Medical Research, Kitchener, Ontario
  - Mor Urology, Inc., Newmarket, Ontario
  - Dr. Bernard Goldfarb, MD, North Bay, Ontario
  - The Fe/Male Health Centres, Oakville, Ontario
  - Dr. John Mahoney, Ottawa, Ontario
  - Allan Abramovitch, MD, Scarborough Village, Ontario
  - Anthony Skehan Medicine Professional Corp., Thunder Bay, Ontario
  - The Male Health Center, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cetrorelix 78 mg
Started | 528
Completed | 473
Not Completed | 55
Not completed — Adverse Event | 8
Not completed — Lack of Efficacy | 10
Not completed — Withdrawal by Subject | 9
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 8
Not completed — incl/excl criterias did not meet | 19

BASELINE CHARACTERISTICS:
Arm/Group | Cetrorelix 78 mg
Number analyzed (Participants) | 528
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 301
  >=65 years | 227
Age Continuous [Mean (Standard Deviation); unit: years] | 64.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 528
Region of Enrollment [Number; unit: participants]
  United States | 414
  Canada | 114

OUTCOME MEASURES:

1. Primary Outcome: IPSS Change From Baseline
Description: International Prostate Symptom Score (IPSS) Patient Questionnaire assessing 7 items (incomplete voiding, frequency, intermittency, urgency, weak stream, hesitancy, nocturia) on a scale from 0 (best) to 5 (worst); total range: 0 - 35 points; absolute change from baseline to Week 26
Time Frame: Baseline and Week 26
Population: Intention to treat (ITT) analysis with Last Observation Carried Forward (LOCF) imputation technique
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cetrorelix 78 mg
Number analyzed (Participants) | 528
Units on a scale | -5.6 (7.1)
Statistical Analysis 1: Comparison: Cetrorelix 78 mg; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -5.6, Standard Deviation 7.1

ADVERSE EVENTS:
Arm/Group | Cetrorelix 78 mg
Serious Adverse Events (participants affected / at risk) | 12/528
Other Adverse Events (participants affected / at risk) | 49/528
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetrorelix 78 mg (N=528)
appendicitis (Infections and infestations) | 1
substance abuse (Psychiatric disorders) | 1
hemorrhagic stroke (Vascular disorders) | 1
chest pain (Cardiac disorders) | 1
coronary artery disease (Cardiac disorders) | 1
rectal abcess (Infections and infestations) | 1
humerus fracture (Injury, poisoning and procedural complications) | 1
bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
chest discomfort (Cardiac disorders) | 1
chest pain / elevated cardiac enzymes (Cardiac disorders) | 1
peripheral artery anuerysm / aortic aneurysm (Vascular disorders) | 1
small intestinal obstruction (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetrorelix 78 mg (N=528)
Hot flush (Vascular disorders) | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less